CLINICAL TRIAL: NCT00517179
Title: Effect of Vardenafil on Blood Pressure in Patients With Erectile Dysfunction Who Received Concomitant Doxazosin GITS for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Effect of Vardenafil on Blood Pressure in Patients With Erectile Dysfunction Who Received Concomitant Doxazosin GITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRE-2006.017-T; HARECCTR0500057
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Prostatic Hyperplasia; Impotence
Keywords: Benign Prostatic Hyperplasia (BPH); Erectile Dysfunction (ED)
MeSH Terms: conditions — Prostatic Hyperplasia; Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

INTERVENTIONS:
Drug: Vardenafil 10mg

SUMMARY:
The purpose of this study is to investigate the interaction between doxazosin GITS and vardenafil on blood pressure (Both systolic and diastolic blood pressure) in patients with both ED and BPH.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 to 80 years old
* Clinically diagnosed to have lower urinary tract symptoms secondary to BPH:

  1. Suffered from lower urinary tract symptoms with International Prostate Symptom Score (IPSS) >=8
  2. Detectable prostatic enlargement determined by Digital Rectum Examination (DRE)
  3. Urinary flow between 5 to 15ml/second in a total void volume >=150mL
* Currently on regular doxazosin GITS once-daily for at least 4 weeks without clinically significant side effects
* Complaints of erectile dysfunction with Erectile Function domain (EF) of the International Index of Erectile Function (IIEF) score <= 21

Exclusion Criteria:

* Congestive heart failure, unstable angina, arrhythmia, myocardial infraction
* Hypertension or on any antihypertensive agents
* Take nitrate and medication contradicted to vardenafil
* Uncontrolled or poorly controlled diabetes mellitus
* Intolerance or contra-indicated for the use of vardenafil
* Hepatic disorder

Ages: 50 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-04; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Mean maximal change of the standing systolic blood pressure (SBP) from half hour prior to till six hour after administration of the drug (baseline) with vardenafil administration versus placebo | From half hour prior to till six hour after administration of the drug (baseline)

SECONDARY OUTCOMES:
Mean maximal post-baseline change of the standing and supine diastolic blood pressure (DBP) | From half hour prior to till six hour after administration of the drug (baseline)
Mean maximal post-baseline change supine SBP, and (3) the pattern of changes of the SBP and DBP from half hour prior to till six hours after administration of the drug | From half hour prior to till six hour after administration of the drug (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, Dr, Principal Investigator — Department of Surgery, Division of Urology, The Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China